CLINICAL TRIAL: NCT06473870
Title: Understanding Lung Cancer Related Risk Factors and Their Impact
Acronym: LUCIA
Status: Not yet recruiting | Type: Observational
Sponsor: Biobizkaia Health Research Institute (Other Government)
Collaborators: Technion, Israel Institute of Technology (Other); Centro Nacional de Análisis Genómico (Unknown); Vicomtech (Unknown); University of Latvia (Other); Centre Hospitalier Universitaire de Liege (Other); Andaluz Health Service (Other Government); Nanose Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LUCIA
Record Dates: First submitted 2024-05-16; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer Screening
Keywords: Lung Cancer; Lung cancer screening; LDCT; Risk factors
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood samples for DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Adult subjects (40 years old or higher), smokers and non-smokers, both women and men who have the capacity to comply with the study follow-up and sign the informed consent, will be recruited from "Servicio Andaluz de Salud" (SAS), "Osakidetza Servicio Vasco de Salud" (OSA), "Centre Hospitalier Universitaire de Liège" (CHUL) and "Centre for Tuberculosis and Lung Diseases (CTLD) of Riga East University Hospital (REUH)".

SUMMARY:
LUCIA aims to develop prediction models for the early diagnosis of lung cancer based on the identification of risk factors and deeper cellular knowledge, by recording real-world data; with risk assessment tools, non-invasive devices and omics analysis. These models will enable new clinical pathways and diagnostic workflow to be implemented to ensure early diagnosis and confirmation, including classification of lung cancer subtype.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death worldwide, causing more deaths than breast and prostate cancer combined.

The current five-year survival rate after diagnosis of all types of lung cancer in Europe is 13% (11.2% for men and 13.9% for women). The five-year survival rate for some types of lung cancer ranges from 6% to 7% (small cell LC) and 23% to 28% for non-small cell lung cancer (NSCLC).

Currently there are important deficiencies when it comes to achieving an adequate lung cancer screening program. According to principles established in 1968, a screening program should be based on pathology that can be improved through the use of population screening.

The evidence suggests two important gaps in early detection. On the one hand, the identification of risk factors beyond smoking and age. And on the other hand, the only tool for early detection that has been shown to reduce morbidity and mortality in lung cancer is chest CT, a test that may not be sustainable in the long term for many healthcare systems. In parallel, lung cancer diagnoses among never smokers and reduced smokers are increasing rapidly, suggesting that if lung cancer screening research continues focusing only on the heaviest smokers, a gap will persist between the population that performs the test and the population that suffers from the disease.

Evidence also suggests that people undergoing screening are not being optimally referred for follow-up or kept engaged in long-term screening.

Currently there are important deficiencies when it comes to achieving an adequate lung cancer screening program. The incidence in individuals without a history of smoking is increasingly higher. Therefore, an observational, longitudinal, multicenter cohort analytical study will be conducted to determine eligibility for screening based on individualized risk (based on age, a more detailed smoking history, occupational exposure, and other risk factors such as ethnicity and family history of lung cancer) and the development and validation of lung cancer risk predictive models that can improve screening efficiency and reduce lung cancer morbidity and mortality.

These models will allow new clinical pathways and diagnostic workflow to be implemented to ensure rapid diagnosis and confirmation, including lung cancer subtype classification.

The study consists of collecting data from participants in 4 visits over two years. During each visit, the clinical evaluation will be carried out, which will consist of the collection of sociodemographic data and clinical history, physical examination, concomitant medication, collection of exposure data and guide symptoms, Quality of Life questionnaires and geolocation. In addition, the following tests will be performed: low-dose computed tomography (LDCT), blood tests, genomic analysis and tests with new non-invasive devices (spectrometry on card (SPOC), breath analyzer (BAN) and broad-spectrum biomarker sensor patch (WBSP)). With all this, the aim is to develop and validate new tests based on new non-invasive and easy-to-use technologies that allow for the implementation of more efficient, acceptable and equitable population screening programs in the near future.

The completion of this project will allow to provide data that can be used to better understand and discover new risk factors for suffering from lung cancer and therefore improve the management of the disease.

Furthermore, this study will favor the reduction of long-term morbidity and mortality from lung cancer and will allow the future implementation of a lung cancer program.

ELIGIBILITY:
Inclusion Criteria (for the 3 phases):

* Subjects aged between 40 and 80 years
* Both genders, of which at least 37% must be women to ensure representativeness
* Willingness and ability to comply with scheduled visits, laboratory tests, and other trial procedures
* Written informed consent obtained prior to performing any protocol-related procedures.

Inclusion criteria for Phase 2: Precision Screening:

* High risk of developing Lung Cancer volunteers will be selected by Lung Cancer risk factors modelling.

Inclusion criteria for Phase 3: Diagnosis:

- Patients diagnosed with indeterminate pulmonary nodules or Lung Cancer from the screening phases.

Exclusion Criteria:

* Subjects under 40 years of age
* Unable to be followed-up for at least 2-years or complete the study
* Subjects that do not sign the informed consent
* Current or prior history of lung cancer
* History of neoplasia in the previous 5 years except non-melanoma skin cancer
* Moderate-severe comorbidities that prevent completion of a diagnostic study in the event of findings suggestive of lung neoplasia (by means of the investigator's clinical judgment) or surgical intervention (< 6 months) if not previously confirmed by cytohistology.
* Vulnerable subjects: severe psychiatric comorbidity, adults under guardianship or deprived of liberty
* Pregnant women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects (40 years old or higher), smokers and non-smokers, both women and men who have the capacity to comply with the study follow-up and sign the informed consent, will be recruited from "Servicio Andaluz de Salud" (SAS), "Osakidetza Servicio Vasco de Salud" (OSA), "Centre Hospitalier Universitaire de Liège" (CHUL) and "Centre for Tuberculosis and Lung Diseases (CTLD) of Riga East University Hospital (REUH)".
Sampling Method: Non-Probability Sample
Enrollment: 6160 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
presence of pulmonary nodules | 2 years
  The main variable is the presence of pulmonary nodules identified by Low Dose Computerized Tomography (LDCT)
Lung Cancer diagnosis | 2 years
  The main variable is the presence of Lung Cancer diagnosis identified by Low Dose Computerized Tomography (LDCT).

SECONDARY OUTCOMES:
Age | 2 years
  years
Gender | 2 years
  Male/female
Ethnicity | 2 years
  description of the ethnia
Socioeconomic factors | 2 years
  deprivation index
Education level | 2 years
  description of the education level
height | 2 years
  meter
weight | 2 years
  kilograms
Body Mass Index | 2 years
  kg/m^2
Blood pressure | 2 years
  Systolic and diastolic blood pressure in mmHg
heart rate | 2 years
  beats/min
respiratory rate | 2 years
  breaths/min
Global Initiative for Obstructive Lung Disease (GOLD) classification | 2 years
  only for COPD patient classification. Grade: GOLD 1 to 4 (from GOLD 1 which means mild stage of COPD to GOLD 4 very severe stage of COPD) Exacerbation history: GOLD A, B or E (depending on exacerbations: Gold A id 0 or 1 moderate exacerbations (not leading to hospitalization) with mMRC 0-1 CAT<10; GOLD B if 0 or 1 moderate exacerbations (not leading to hospitalization) with mMRC >= 2 CAT >=10 and GOLD E if 2 or more moderate exacerbations or 1 or more leading to hospitalization) with mMRC 0-1 CAT<10.
Medical record | 2 years
  Family history of lung cancer or other types of cancer, emphysema/ COPD (+ GOLD classification)/ asthma, Interstitial Lung Disease (interstitial patterns), bronchiectasis, arterial hypertension, dyslipidemia, previous acute myocardial infarction, vasculopathies and chronic treatment.
Exposure to harmful agents | 2 years
  Smoking and occupational exposure (physical activity and frequency, alcohol intake, cigarette packets/year, age of smoking onset, time elapsed since last cigarette, occupational exposure to carcinogens).
Exploratory Omics markers | baseline
  Dedicated blood samples will be specifically performed for a large Omics analysis.
HEALTH-PROMOTING LIFESTYLE PROFILE II questionnaire (HPLP II) | 2 years
  A score for overall health-promoting lifestyle is obtained by calculating a mean of the individual's responses to all 52 items; six subscale scores are obtained similarly by calculating a mean of the responses to subscale items. The use of means rather than sums of scale items is recommended to retain the 1 to 4 metric of item responses and to allow meaningful comparisons of scores across subscales.
  Lower scores (1) mean lower engage in a health-promoting lifestyle Higher scores (4) mean higher engage in a health-promoting lifestyle
Fantastic lifestyle Checklist | 2 years
  Evaluation of the population lifestyle:
  85-100 points --> Excellent 70-84 points --> Very good 55-69 points --> Good 35-54 points --> Fair 0-34 points --> needs improvement
Mediterranean diet adherence questionnaire | 2 years
  0-14 points scale <9 points --> low adherence to Mediterranean diet >9 points --> High adherence to Mediterranean diet
EuroQoL-5D-5L questionnaire | 2 years
  Scoring from 0-100 points. 0 points low quality of life 100 high quality of life
The Alcohol Use Disorders Identification Test (AUDIT) questionnaire | 2 years
  Scoring from 0-40 points >8 points --> indicators of hazardous and harmful alcohol use 8-15 points --> simple advice focused on the reduction of hazardous drinking 16-19 points --> brief counseling and continued monitoring >20 points --> warrant further diagnostic evaluationfor alcohol dependence
Breath Analyzer (BAN) device | 2 years
  Measurement of Volatile Organic Compounds (VOCs) of a breath sample for Lung Cancer early detection
Wide-biomarker-spectrum Multi-Use Sensing Patch (WBSP) | 2 years
  Measurement of Volatile Organic Compounds (VOCs) in the sweat and skin headspace for Lung Cancer early detection
Spectrometry-on-Card (SPOC) | 2 years
  Measurement of biomarkers and signals from a blood sample for the early detection of lung cancer
Tumor pathology | 2 years
  Tumor biopsy will be carried out in order to classify and characterize it regarding its size and location.
Lung CT scan description | 2 years
  A lungCT scan will be performed to. Lung nodules and other findings (if any) will be reported in order to diagnose a lung cancer. If no anomalies are found, it will also be reported.
Forced Vital Capacity (FVC) | 2 years
  mL, %, Lower limit of Normal and z-score
Forced Expiratory Volume in 1 second (FEV1) | 2 years
  mL, %, Lower limit of Normal and z-score
FEV1/FVC ratio | 2 years
  percentage (%)
Glucose | baseline
  mg/dL
HDL Cholesterol | baseline
  mg/dL
Iron | baseline
  μg/dL
C reactive protein | baseline
  mg/L
Proteins | baseline
  g/dL
Albumin | baseline
  g/dL
LDL Cholesterol | baseline
  mg/dL
Ferritin | baseline
  ng/mL
Chloride | baseline
  mEq/L
Lactate dehydrogenase | baseline
  U/L
Triglycerides | baseline
  mg/dL
Transferrin Index | baseline
  index
Cholesterol | baseline
  mg/dL
transferrin | baseline
  mg/dL
phosphate | baseline
  mg/dL
calcium | baseline
  mg/dL
GOT | baseline
  U/L
GPT | baseline
  U/L
GGT | baseline
  U/L
Bilirubin | baseline
  mg/dL
Alkaline phosphatase | baseline
  U/L
urea | baseline
  mg/dL
Creatinine | baseline
  mg/dL
Sodium | baseline
  mEq/L
potassium | baseline
  mEq/L
Urate | baseline
  mg/dL
carcinoembryonic antigen (CEA) | baseline
  ng/mL
CA 125 | baseline
  U/mL
CYFRA 21.1 | baseline
  ng/mL
Neuronal specific enolase (NSE) | baseline
  ng/mL
Complete blood count | baseline
  number of blood cells, composition and percentage
erythrocyte sedimentation rate | baseline
  mm/h
partial thromboplastin time | baseline
  seg
fibrinogen | baseline
  mg/dL
international normalized ratio (INR) | baseline
  ratio
prothrombin time | baseline
  seg
Geo location | 2 years
  Participant's census tract identification (one for home address and one for workplace address)

CONTACTS AND LOCATIONS:
Overall Officials: Luis G Luque-Romero, MD, Principal Investigator — Andaluz Health Service; David Vicente-Baz, MD, Principal Investigator — Andaluz Health Service; Alvils Krams, MD, Principal Investigator — University of Latvia; Julien Guiot, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (5):
- Centre Hospitalier Universitaire de Liège, Liège, Wallonia, Belgium
- Riga East University Hospital, Riga, Latvia
- Spain (3):
  - Hospital Universitario Cruces, Barakaldo, Viscay
  - Hospital Universitario Virgen Macarena, Seville
  - Aljarafe-Sevilla Norte Health District, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Meerbeeck JP, Franck C. Lung cancer screening in Europe: where are we in 2021? Transl Lung Cancer Res. 2021 May;10(5):2407-2417. doi: 10.21037/tlcr-20-890. PMID 34164288
- [Background] Oudkerk M, Liu S, Heuvelmans MA, Walter JE, Field JK. Lung cancer LDCT screening and mortality reduction - evidence, pitfalls and future perspectives. Nat Rev Clin Oncol. 2021 Mar;18(3):135-151. doi: 10.1038/s41571-020-00432-6. Epub 2020 Oct 12. PMID 33046839
- [Background] Adams SJ, Stone E, Baldwin DR, Vliegenthart R, Lee P, Fintelmann FJ. Lung cancer screening. Lancet. 2023 Feb 4;401(10374):390-408. doi: 10.1016/S0140-6736(22)01694-4. Epub 2022 Dec 20. PMID 36563698
- [Background] Gomez-Carballo N, Fernandez-Soberon S, Rejas-Gutierrez J. Cost-effectiveness analysis of a lung cancer screening programme in Spain. Eur J Cancer Prev. 2022 May 1;31(3):235-244. doi: 10.1097/CEJ.0000000000000700. PMID 34406177
- [Background] Thandra KC, Barsouk A, Saginala K, Aluru JS, Barsouk A. Epidemiology of lung cancer. Contemp Oncol (Pozn). 2021;25(1):45-52. doi: 10.5114/wo.2021.103829. Epub 2021 Feb 23. PMID 33911981
- [Background] Schabath MB, Cote ML. Cancer Progress and Priorities: Lung Cancer. Cancer Epidemiol Biomarkers Prev. 2019 Oct;28(10):1563-1579. doi: 10.1158/1055-9965.EPI-19-0221. PMID 31575553
- [Background] Zhang T, Joubert P, Ansari-Pour N, Zhao W, Hoang PH, Lokanga R, Moye AL, Rosenbaum J, Gonzalez-Perez A, Martinez-Jimenez F, Castro A, Muscarella LA, Hofman P, Consonni D, Pesatori AC, Kebede M, Li M, Gould Rothberg BE, Peneva I, Schabath MB, Poeta ML, Costantini M, Hirsch D, Heselmeyer-Haddad K, Hutchinson A, Olanich M, Lawrence SM, Lenz P, Duggan M, Bhawsar PMS, Sang J, Kim J, Mendoza L, Saini N, Klimczak LJ, Islam SMA, Otlu B, Khandekar A, Cole N, Stewart DR, Choi J, Brown KM, Caporaso NE, Wilson SH, Pommier Y, Lan Q, Rothman N, Almeida JS, Carter H, Ried T, Kim CF, Lopez-Bigas N, Garcia-Closas M, Shi J, Bosse Y, Zhu B, Gordenin DA, Alexandrov LB, Chanock SJ, Wedge DC, Landi MT. Genomic and evolutionary classification of lung cancer in never smokers. Nat Genet. 2021 Sep;53(9):1348-1359. doi: 10.1038/s41588-021-00920-0. Epub 2021 Sep 6. PMID 34493867
- [Background] Ramaswamy A. Lung Cancer Screening: Review and 2021 Update. Curr Pulmonol Rep. 2022;11(1):15-28. doi: 10.1007/s13665-021-00283-1. Epub 2022 Apr 2. PMID 35402145
- [Background] Ten Haaf K, van der Aalst CM, de Koning HJ, Kaaks R, Tammemagi MC. Personalising lung cancer screening: An overview of risk-stratification opportunities and challenges. Int J Cancer. 2021 Jul 15;149(2):250-263. doi: 10.1002/ijc.33578. Epub 2021 May 3. PMID 33783822
- [Background] Berghmans T, Lievens Y, Aapro M, Baird AM, Beishon M, Calabrese F, Degi C, Delgado Bolton RC, Gaga M, Lovey J, Luciani A, Pereira P, Prosch H, Saar M, Shackcloth M, Tabak-Houwaard G, Costa A, Poortmans P. European Cancer Organisation Essential Requirements for Quality Cancer Care (ERQCC): Lung cancer. Lung Cancer. 2020 Dec;150:221-239. doi: 10.1016/j.lungcan.2020.08.017. Epub 2020 Sep 4. PMID 33227525
- [Background] Lemjabbar-Alaoui H, Hassan OU, Yang YW, Buchanan P. Lung cancer: Biology and treatment options. Biochim Biophys Acta. 2015 Dec;1856(2):189-210. doi: 10.1016/j.bbcan.2015.08.002. Epub 2015 Aug 19. PMID 26297204
- [Background] Nasim F, Sabath BF, Eapen GA. Lung Cancer. Med Clin North Am. 2019 May;103(3):463-473. doi: 10.1016/j.mcna.2018.12.006. PMID 30955514
- [Background] Nooreldeen R, Bach H. Current and Future Development in Lung Cancer Diagnosis. Int J Mol Sci. 2021 Aug 12;22(16):8661. doi: 10.3390/ijms22168661. PMID 34445366
- [Background] Liu Y, Pan IE, Tak HJ, Vlahos I, Volk R, Shih YT. Assessment of Uptake Appropriateness of Computed Tomography for Lung Cancer Screening According to Patients Meeting Eligibility Criteria of the US Preventive Services Task Force. JAMA Netw Open. 2022 Nov 1;5(11):e2243163. doi: 10.1001/jamanetworkopen.2022.43163. PMID 36409492
- [Background] Braithwaite D, Gould MK. Is Lung Cancer Screening Reaching the People Who Are Most Likely to Benefit? JAMA Netw Open. 2022 Nov 1;5(11):e2243171. doi: 10.1001/jamanetworkopen.2022.43171. No abstract available. PMID 36409500
- [Background] Ten Haaf K, Jeon J, Tammemagi MC, Han SS, Kong CY, Plevritis SK, Feuer EJ, de Koning HJ, Steyerberg EW, Meza R. Risk prediction models for selection of lung cancer screening candidates: A retrospective validation study. PLoS Med. 2017 Apr 4;14(4):e1002277. doi: 10.1371/journal.pmed.1002277. eCollection 2017 Apr. PMID 28376113
- [Background] Gould MK, Huang BZ, Tammemagi MC, Kinar Y, Shiff R. Machine Learning for Early Lung Cancer Identification Using Routine Clinical and Laboratory Data. Am J Respir Crit Care Med. 2021 Aug 15;204(4):445-453. doi: 10.1164/rccm.202007-2791OC. PMID 33823116
- [Background] Yeh MC, Wang YH, Yang HC, Bai KJ, Wang HH, Li YJ. Artificial Intelligence-Based Prediction of Lung Cancer Risk Using Nonimaging Electronic Medical Records: Deep Learning Approach. J Med Internet Res. 2021 Aug 3;23(8):e26256. doi: 10.2196/26256. PMID 34342588
- [Background] de Koning HJ, van der Aalst CM, de Jong PA, Scholten ET, Nackaerts K, Heuvelmans MA, Lammers JJ, Weenink C, Yousaf-Khan U, Horeweg N, van 't Westeinde S, Prokop M, Mali WP, Mohamed Hoesein FAA, van Ooijen PMA, Aerts JGJV, den Bakker MA, Thunnissen E, Verschakelen J, Vliegenthart R, Walter JE, Ten Haaf K, Groen HJM, Oudkerk M. Reduced Lung-Cancer Mortality with Volume CT Screening in a Randomized Trial. N Engl J Med. 2020 Feb 6;382(6):503-513. doi: 10.1056/NEJMoa1911793. Epub 2020 Jan 29. PMID 31995683
- [Background] US Preventive Services Task Force; Krist AH, Davidson KW, Mangione CM, Barry MJ, Cabana M, Caughey AB, Davis EM, Donahue KE, Doubeni CA, Kubik M, Landefeld CS, Li L, Ogedegbe G, Owens DK, Pbert L, Silverstein M, Stevermer J, Tseng CW, Wong JB. Screening for Lung Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2021 Mar 9;325(10):962-970. doi: 10.1001/jama.2021.1117. PMID 33687470
- [Background] Triplette M, Wenger DS, Shahrir S, Kross EK, Kava C, Phipps A, Hawes SE, Cole A, Snidarich M, Crothers K. Patient Identification of Lung Cancer Screening Follow-Up Recommendations and the Association with Adherence. Ann Am Thorac Soc. 2022 May;19(5):799-806. doi: 10.1513/AnnalsATS.202107-887OC. PMID 34727513
- [Background] Lin Y, Fu M, Ding R, Inoue K, Jeon CY, Hsu W, Aberle DR, Prosper AE. Patient Adherence to Lung CT Screening Reporting & Data System-Recommended Screening Intervals in the United States: A Systematic Review and Meta-Analysis. J Thorac Oncol. 2022 Jan;17(1):38-55. doi: 10.1016/j.jtho.2021.09.013. Epub 2021 Oct 6. PMID 34624528
- [Background] Rivera GA, Wakelee H. Lung Cancer in Never Smokers. Adv Exp Med Biol. 2016;893:43-57. doi: 10.1007/978-3-319-24223-1_3. PMID 26667338
- [Background] Smith RJ, Vijayaharan T, Linehan V, Sun Z, Ein Yong JH, Harris S, Mariathas HH, Bhatia R. Efficacy of Risk Prediction Models and Thresholds to Select Patients for Lung Cancer Screening. Can Assoc Radiol J. 2022 Nov;73(4):672-679. doi: 10.1177/08465371221089899. Epub 2022 Apr 26. PMID 35471946
- [Background] Tammemagi MC, Ten Haaf K, Toumazis I, Kong CY, Han SS, Jeon J, Commins J, Riley T, Meza R. Development and Validation of a Multivariable Lung Cancer Risk Prediction Model That Includes Low-Dose Computed Tomography Screening Results: A Secondary Analysis of Data From the National Lung Screening Trial. JAMA Netw Open. 2019 Mar 1;2(3):e190204. doi: 10.1001/jamanetworkopen.2019.0204. PMID 30821827
- See also: Lung Cancer Survival Rates — http://www.cancer.org/cancer/lung-cancer/detection-diagnosis-staging/survival-rates.html
- See also: GLOBOCAN 2020: Estimated cancer incidence, mortality and prevalence worldwide in 2020 — http://gco.iarc.fr/today/data/factsheets/populations/900-world-fact-sheets.pdf
- See also: Proposal for a Council Recommendation on strengthening prevention through early detection: A new EU approach on cancer screening replacing Council Recommendation 2003/878/EC — http://eur-lex.europa.eu/legal-content/EN/TXT/?uri=CELEX%3A52022SC0296&qid=1664222001392